CLINICAL TRIAL: NCT04260490
Title: Multiple Myeloma in the French West Indies. Environmental and Professional Exposure to Pesticide: A Case-control Study in Guadeloupe and Martinique
Brief Title: Multiple Myeloma and Environmental Exposure to Pesticides in the French West Indies: A Population Based Case-control Study.
Acronym: MYELODOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Guadeloupe Cancer Registry (Unknown); Martinique Cancer Registry (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Liege (Other); University Hospital Center of Martinique (Other); Centre Hospitalier de Basse-Terre (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAP_RI2_2018/01
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; pesticide; chlordecone; Guadeloupe; Martinique
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma collection and DNA collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases will be interviewed using a standardized questionnaire. Blood samples will be taken for standard and specific analyses. Samples for chlordecone and other Persistent organic Polluants (POPs) tests will be collected.
  Blood samples will be collected for the biobank of Guadeloupe for further studies on genetic susceptibility markers and their links with pesticide exposure.
- Controls: Controls selected after stratification on department of residence, sex and age of the cases and who give a written informed consent to participate.
  Controls will be interviewed using a standardized questionnaire. Blood samples will be taken for standard and specific analyses in both cases and controls. Samples for chlordecone and other Persistent organic Polluants (POPs) tests will be collected. Blood samples will be collected for the biobank of Guadeloupe for further studies on genetic susceptibility markers and their links with pesticide exposure.

SUMMARY:
Multiple myeloma (MM) is a malignancy of plasma cells engaging in monoclonal immunoglobulin production. A strong presumption was established between exposure to pesticides and the risk of MM. The French West Indies departments of Guadeloupe and Martinique are characterized by a wide use of pesticides related to bananas plantation, particularly chlordecone which has been classified by IARC as possibly carcinogenic and has recognized hormonal properties (endocrine disruptor). The objective of this study is to measure the association between exposure to pesticide and other environmental factors in the occurrence of MM in Guadeloupe and Martinique and to estimate the proportion of cases of MM attributable to pesticide exposure. Genetic susceptibility markers and their links to environmental factors will be subsequently studies from blood samples collection.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a mature B-cell lymphoma characterized by monoclonal proliferation of tumor plasma cells invading the bone marrow. It is the second malignant hemopathy among Non-Hodgkin's Lymphomas. Etiology of the disease is poorly understood. Its higher incidence in black subjects suggests the existence of genetic factors. Numerous studies have evoked the role of exposure to environmental and occupational factors in the occurrence of MM such as exposure to pesticides, solvents, in particular benzene, and other petroleum derivatives, as well as work in an agricultural environment, in hairdressing and in the metallurgical and textile industries. According to the Collective Inserm expertise "Pesticides and Health", a strong presumption (++) has been established between exposure to pesticides and the risk of occurrence of MM.

In the French West Indies (Guadeloupe, Martinique), the incidence of MM is higher than in France. These 2 departments are characterized by a major use of pesticides in connection with the banana culture developed intensively from the 1950s. These cultures successively used organochlorine insecticides, mainly β-hexachlorocyclohexane (β-HCH), technical HCH (mixture of α, β, and γ isomers of HCH), and especially chlordecone (CLD). CLD was used from 1972 to 1993 under the trade names of Kepone® (1972-1978) and then Curlone® (1982-1993) with a CLD rate of 5%. The absence of biotic and abiotic degradation of CLD has resulted in persistent soil pollution, still present today, contamination of surface and deep waters, many plant and animal products, terrestrial and marine, and then the population. CLD is a proven carcinogen in rodents, classified as a possible carcinogen by the International Agency for Research on Cancer (IARC) and has recognized hormonal properties (endocrine disruptor). CLD has been associated with an increased risk of prostate cancer in Guadeloupe. In Martinique, a geographic correlation study has shown a high incidence of MM in individuals residing on soils polluted by CLD.

Studies on the impact of pesticides on health come up against numerous limits, in the foreground of which is the great diversity of products (more than 900 active ingredients were approved one day in France and marketed in more than 9000 different products) and the difficulty in reconstructing retrospectively and objectively the exposures of individuals due to the multiplicity of sources of exposure (leisure, gardening, domestic use).

Mode of action of pesticides is still insufficiently documented, but some are classified as genotoxic, immunotoxic, tumor promoters or endocrine disruptors. Data available in the literature mainly relate to case-control or cohort studies on the occupational exposure of agricultural workers in industrialized countries. Measurement of this exposure is mainly made from self-administered questionnaires.

The investigators propose to assess feasibility of a case-control study on role of exposure to pesticides, in particular to CLD and persistent pollutants, as well as other occupational exposures in the occurrence of MM in the West Indies. This study is part of the recommendations of the Inserm-InVs Chlordecone Scientific Council and action 18 of the National Interministerial Chlordecone Plan "initiate work on the link between myelomas and exposure to chlordecone".

ELIGIBILITY:
Inclusion Criteria:

* Cases :
* patients above 18 years old
* with a place of residence in Guadeloupe or Martinique
* meeting the inclusion criteria for multiple myeloma identified from hematologist, oncologist and clinicians
* who ave a written informed consent.

Controls :

* individuals selected after stratification on department of residence, sex and age of the cases
* who gave a written informed consent to participate.

Exclusion Criteria:

* Refusal to participate
* subject not affiliated to a social welfare or under guardianship
* Pregnant or lactating woman
* Subject participating in another research including an exclusion period still in progress at the pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A case-control study in the general population with etiological aim, paired multicentric will be carried out. This choice is justified given the low frequency of the pathology studied in the two islands.
  Cancer registries of Guadeloupe and Martinique exhaustively collect cases of multiple myeloma (MM) according to cancer registration rules established at European and international level. They have data to identify the usual places of care and diagnosis of MM in their respective territory and work in close collaboration with clinical services in charge of patients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Measure of association between exposure to chlordecone and risk of multiple myeloma. | Pesticide samples will be sent to the Reference Laboratory of Animal Ecology and Ecotoxicology in Liège once or twice a year. For a given patient, the time frame (questionnaire + and blood analyses) will be 12 months after inclusion.
  The exposure measurement will be done using several complementary methods combining:
  * Serum dosages of chlordecone + Persistent Organic Pollutant
  * Evaluation from questionnaires
  * Use of job-exposure matrices (benzene and other solvents), made available by the Occupational Health Department (DST) of the Institute for Health Monitoring (InVS)
  * Use of crop-exposure matrices : the banana crop matrix developed for the Antilles by the DST of InVS in collaboration with the Interregional Epidemiology Unit (CIRE) Antilles Guyane and will be used

SECONDARY OUTCOMES:
proportion of MM cases attributable to pesticide exposure | 36 months after first inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Deloumeaux, MD, Principal Investigator — CHU de la Guadeloupe
Locations (2):
- University Hospital Center of Guadeloupe, Pointe-à-Pitre, Guadeloupe
- University Hospital Center of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flowers CR, Glover R, Lonial S, Brawley OW. Racial differences in the incidence and outcomes for patients with hematological malignancies. Curr Probl Cancer. 2007 May-Jun;31(3):182-201. doi: 10.1016/j.currproblcancer.2007.01.005. No abstract available. PMID 17543947
- [Background] Multigner L, Ndong JR, Giusti A, Romana M, Delacroix-Maillard H, Cordier S, Jegou B, Thome JP, Blanchet P. Chlordecone exposure and risk of prostate cancer. J Clin Oncol. 2010 Jul 20;28(21):3457-62. doi: 10.1200/JCO.2009.27.2153. Epub 2010 Jun 21. PMID 20566993